CLINICAL TRIAL: NCT01790009
Title: Influence of Age on the Absorption and Metabolism of Cocoa Flavanols
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Reading (Other)
Responsible Party: Principal Investigator, Jeremy Paul Edward Spencer, Professor, University of Reading
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FLAV-AGE01
Record Dates: First submitted 2013-02-08; First posted 2013-02-12 (Estimated); Last update posted 2013-02-12 (Estimated); Status verified 2013-02

CONDITIONS: Healthy
Keywords: ADME; Flavanols; Age; Pharmacokinetics
MeSH Terms: interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Flavanol Rich drink (Active Comparator): Flavanol-rich drink containing 800 mg/75 Kg of Body Weight (BW)
  Interventions: Dietary Supplement: Flavanol rich drink
- Flavanol rich drink (Active Comparator): Flavanol Intervention drink 400 mg/75 Kg BW
  Interventions: Dietary Supplement: Flavanol rich drink
- Acetaminophen (Active Comparator): 2 tabletsx500 mg
  Interventions: Drug: Acetaminophen

INTERVENTIONS:
Dietary Supplement: Flavanol rich drink
  Other Names: Comparison of two different doses of a flavanol rich drink
  Arms: Flavanol Rich drink; Flavanol rich drink
Drug: Acetaminophen — 2x500 mg Acetaminophen
  Other Names: Paracetamol
  Arms: Acetaminophen

SUMMARY:
Accumulating evidence suggests that regular consumption of foods and beverages rich in flavanols, such as cocoa, tea, apples and wine, may have cardiovascular benefits. Several well-controlled randomised human intervention studies have shown that cocoa flavanols have beneficial effects on blood pressure, endothelial function and other biomarkers of cardiovascular health. These vascular improvements have been correlated in time with changes in plasma flavanol metabolites. The health benefits of flavanol consumption are therefore likely dependent on changes in their absorption, distribution, metabolism and excretion (ADME). Recent studies have provided detailed information regarding the absorption and metabolism of cocoa flavanols. However, there is a lack of information on whether there are changes in flavanol absorption and metabolism with increasing age.

ELIGIBILITY:
Inclusion Criteria:

* signed consent form
* Caucasian
* Good general health
* No allergy to milk products or sensitivity to alkaloids/caffeine,
* No gastrointestinal disorders (e.g., chronic constipation, diarrhoea, inflammatory bowel disease, irritable bowel syndrome, or other chronic gastrointestinal complaints)
* Not diabetic or suffering from hypertension (140/90 mm Hg),
* No anaemia or gall bladder problems.

Exclusion Criteria:

* those on a weight reducing dietary regimen
* Taking any dietary supplements
* Consuming more than 15 units (120g) of alcohol per week
* Taking anti-inflammatory medication
* Smokers
* Those with sensitivities to chocolate, reduced calorie sweeteners, dairy, nuts or gluten,
* Vegetarians or vegans.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-02; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Plasma and urine flavanol metabolites | 24 hours

SECONDARY OUTCOMES:
Paracetamol and methylxanthine plasma and urine levels | 24 h

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Spencer, PhD, Study Director — University of Reading
Locations (1):
- Department of Food and Nutritional Sciences, Reading, Berkshire, United Kingdom